CLINICAL TRIAL: NCT03954652
Title: Whole Genome Trio Sequencing as a Standard Routine Test in Patients With Rare Diseases - "GENOME FIRST APPROACH"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: WG-Trio01
Record Dates: First submitted 2019-05-09; First posted 2019-05-17 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Rare Diseases; Genetic Predisposition
Keywords: Rare Diseases; Genetic Predisposition; Whole-exome sequencing; WGS-trio analysis; Whole Genome Sequencing (WGS)
MeSH Terms: conditions — Rare Diseases; Genetic Predisposition to Disease

STUDY DESIGN:
Intervention Model Description: Cohort 1: IQ < 70 with and without malformations, syndromic and non-syndromic Cohort 2: Retinitis pigmentosa, achromatopsy, Bardet-Biedl syndrome, Usher syndrome, congenital stationary night blindness, LCA, macula degeneration, rod/ cone dystrophies, opticus atrophy Cohort 3: Rare paediatric solid cancers as melanoma, carcinoma of the gastrointestinal tract, tumours of the salivary gland and pancreatic tumors in children.
  Plus: their respective parents
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Intellectual disability (Other): Genetic: WGS Diagnostic Blood take for genetic diagnostic.
  Interventions: Genetic: WGS-Diagnostic
- Cohort 2 Retinal diseases (Other): Genetic: WGS Diagnostic Blood take for genetic diagnostic.
  Interventions: Genetic: WGS-Diagnostic
- Cohort 3: Rare tumors in childhood (Other): Genetic: WGS Diagnostic Blood take for genetic diagnostic.
  Interventions: Genetic: WGS-Diagnostic

INTERVENTIONS:
Genetic: WGS-Diagnostic — Blood sampling, shot clinical characterization, WGS-based trio sequencing, NGS analysis and other omics analysis (transcriptomics, proteomics, metabolomics), functional cell biology studies (for example in fibroblast cultures), RNA-seq.

SUMMARY:
The GENOME FIRST APPROACH project will enroll patients (n = 450) and their healthy parents with unclear molecular cause of the disease, suspected genetic cause of the disease and the healthy parents of those affected for trio analysis (N in total 1350).

DETAILED DESCRIPTION:
In the GENOME FIRST APPROACH (monocentric, prospective, open-label diagnostic) project, patients with molecularly undiagnosed diseases will diagnostically be analyzed by Whole Genome Sequencing (WGS)-trio analysis. The following questions will be leading the project:

Primary:

• Efficacy of WGS trio analysis in different clinical indications

Secondary:

* Systematically benchmark WGS analysis to detect genetic variations compared to WES and single nucleotide polymorphism (SNP) array analysis,
* Expand the analysis from coding single-nucleotide variants (SNVs) to regulatory mutations, structural variants (SVs), and low complexity regions,
* Validate the efficacy of clinical genome trio sequencing in a routine diagnostic setting,
* Analyse whether 42x coverage has the potential to discover mosaicism as disease causing mechanism,
* Further develop algorithms for integrative analyses of Trio-WGS data with Ribonucleic acid- sequencing (RNA-seq),
* Identify de novo alterations and novel disease mechanisms,
* Gain fundamental new insights into disease mechanisms and cellular biology,
* Combine WGS with further Omics methods to improve genetic diagnostics of future rare disease patients, and
* Explore overall financial costs and time to report conclusive data to the patients of the Trio-WGS approach compared to traditional multistep diagnostic approaches using single-gene, panel, whole-exome sequencing (WES) and chromosomal microarray (CMA) (SNP array, array-based comparative genomic hybridization (arrayCGH)) analysis.

In addition, healthy parents of the subjects will be included in the project to perform parent-child (trio) analyzes.

ELIGIBILITY:
Inclusion Criteria:

* Unclear molecular cause of the disease
* Suspected genetic cause of the disease
* Healthy parents of those affected for trio analysis Cohort 1: IQ < 70 with and without malformations, syndromic and non-syndromic Cohort 2: Retinitis pigmentosa, achromatopsy, Bardet-Biedl syndrome, Usher syndrome, congenital stationary night blindness, LCA, macula degeneration, rod/ cone dystrophies, opticus atrophy Cohort 3: Rare paediatric solid cancers as melanoma, carcinoma of the gastrointestinal tract, tumours of the salivary gland and pancreatic tumors in children.

Exclusion Criteria:

Cohort 1: Toxic causes (drugs, infections) Cohort 2: patients with non-genetic forms of blindness Cohort 3: adult cancer, blood cancer

* Missing informed consent of the patient/ legal guardian
* Missing samples of both parents
* Previous WES or panel analysis-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1350 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Full genomic sequence analysis carried out by Whole Genome Sequencing (WGS) | Day 1
  Number of genomic variants in disease and health parents by WGS (a Next-Generation Sequencing Technology, NGS)

SECONDARY OUTCOMES:
Genome sequencing | Day 1
  Verification of the genetic causes of unclear genetic diseases by clinical genome sequencing
De novo alterations | Day 1
  Number of de novo alterations in genome of the enrolled population

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Riess, Prof. Dr., Study Director — University Hospital Tübingen
Locations (1):
- University Hospital Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No